CLINICAL TRIAL: NCT04996030
Title: An Open-label Phase 1 Study to Evaluate Pharmacokinetics, Safety, and Tolerability of SY-2101 in Adult Patients With Acute Promyelocytic Leukemia
Brief Title: A Study for Oral SY-2101 for Participants With Acute Promyelocytic Leukemia
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Prioritization
Sponsor: Syros Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SY-2101-101
Record Dates: First submitted 2021-08-03; First posted 2021-08-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Acute Promyelocytic Leukemia
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide; cyclo-tetrakis(bis(1-phenyl-3-methyl-4-benzoylpyrazolon-5-ato)mu-oxotitanium(IV))

STUDY DESIGN:
Intervention Model Description: The characterization of single-dose PK will be conducted in an open-label, randomized crossover 3-period, 3-treatment, 2-sequence design, separated by ≥1 week of washout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Single-Dose PK Module: Sequence 1 (Experimental): Participants will receive IV ATO in a fasted state on Day 1, SY-2101 in a fed state on Day 8, and SY-210 in a fasted state on Day 15 during Weeks 6, 7, and 8 of any consolidation cycle being received as part of SOC treatment consolidation cycle.
  Interventions: Drug: SY-2101; Drug: Arsenic Trioxide
- Single-Dose PK Module: Sequence 2 (Experimental): Participants will receive IV ATO in a fasted state on Day 1, SY-2101 in a fasted state on Day 8, and SY-2101 in a fed state on Day 15 during Weeks 6, 7, and 8 of any consolidation cycle being received as part of SOC treatment consolidation cycle.
  Interventions: Drug: SY-2101; Drug: Arsenic Trioxide
- Single-Dose PK Comparability Module (Experimental): Participants will receive two single-dose treatments of SY-2101, with separated from one another by approximately 1 week and separated from any preceding IV ATO dose by at least 72 hours.
  Interventions: Drug: SY-2101
- Multiple-Dose IV Module (Experimental): Participants will receive IV ATO, once daily (QD), 5 days/week for 28 days as a part of at least one cycle (Weeks 1 through 4) of SOC treatment consolidation.
  Interventions: Drug: Arsenic Trioxide
- Multiple-Dose Oral Module (Experimental): Participants will receive SY-2101, QD, 5 days/week for 28 days as a part of one cycle (Cycle 4; Weeks 1 through 4) of SOC treatment consolidation.
  Interventions: Drug: SY-2101

INTERVENTIONS:
Drug: SY-2101 — SY-2101 will be administered per dose and schedule specified in arm description.
  Other Names: Oral ATO; Oral Arsenic Trioxide
  Arms: Multiple-Dose Oral Module; Single-Dose PK Comparability Module; Single-Dose PK Module: Sequence 1; Single-Dose PK Module: Sequence 2
Drug: Arsenic Trioxide — IV ATO will be administered per dose and schedule specified in arm description.
  Other Names: IV ATO; Trisenox®; IV Arsenic Trioxide
  Arms: Multiple-Dose IV Module; Single-Dose PK Module: Sequence 1; Single-Dose PK Module: Sequence 2

SUMMARY:
SY-2101 is being studied as a treatment for participants with a type of leukemia called acute promyelocytic leukemia (APL). SY-2101 is an oral formulation of a drug called arsenic trioxide (ATO). ATO is already used to treat APL in a formulation that is given as an intravenous (IV) infusion (through a needle in the arm). SY-2101 is a formulation of ATO that is taken orally (by mouth).

This trial will include participants with APL in remission, who are receiving standard of care (SOC) treatment with all-trans-retinoic acid (ATRA) and IV ATO, during the consolidation phase of chemotherapy or within the past 6 months. The participants in this trial will receive continued treatment with ATO and ATRA to help keep their cancer from coming back. There will be some weeks when participants receive IV ATO and others when they receive SY-2101 (ATO taken orally). Participants with high-risk APL may be eligible for part 1 or 4 of the study for the 6 months following completion of their standard of care ATRA and ATO treatment.

DETAILED DESCRIPTION:
This study includes 4 parts. In the first part, enrolled participants will receive a single dose of IV ATO, followed a week later by a single dose of SY-2101, SY-2101 will be administered to participants in either a fed or a fasted condition. A week after that, participants will receive a second, a single dose of SY-2101, with some participants taking this dose in a fed state and other participants taking this dose in a fasted condition. After each of these doses, blood draws and safety assessments will be performed. In the second part, enrolled participants will receive IV ATO according to the standard of care, with collection of blood and safety assessments. In the third part, enrolled participants who are documented to be in molecular remission will receive SY-2101 in place of IV ATO during the 4th cycle of consolidation, with the collection of blood and safety assessments throughout the cycle. In the fourth part, enrolled participants will receive two single-dose treatments of SY-2101 approximately one week apart.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must have a diagnosis of APL characterized by the presence of the t(15;17) translocation or PML/RARA gene expression via reverse transcription polymerase chain reaction (RT-PCR), fluorescence in situ hybridization (FISH), or cytogenetics. Participants with low-risk APL may be eligible for all parts of this study; participants with high-risk APL are only eligible for the single-dose modules if they have completed a treatment regimen that included ATO within 6 months prior to the Screening Visit.
* Participants must have received ATO plus ATRA induction therapy and must have received or be eligible and planning to receive consolidation therapy with ATO plus ATRA in alignment with National Comprehensive Cancer Network (NCCN) guidelines for low-risk APL prior to their enrollment in the study; or participants must have completed a treatment regimen that included ATO within 6 months prior to the Screening Visit.
* Participants must be able to tolerate full dose ATO per NCCN guidelines.
* Participants must be in morphological complete remission (CR) at the end of induction.
* Participants must have a serum or high-sensitivity urine pregnancy test (for females of childbearing potential) that is negative at the Screening Visit and immediately prior to initiation of study treatment (first dose of study drug).

Key Exclusion Criteria:

* Participants who have demonstrated relapse and therefore are not eligible for further consolidation.
* Participants currently receiving treatment for a non-APL malignancy (not including basal cell carcinoma, non-melanoma skin cancer, cervical carcinoma in situ, or localized prostate cancer treated with hormone therapy). Participants with history of other cancers should be free of disease for at least 2 years prior to the Screening Visit.
* Participants with an active, life-threatening, or clinically-significant uncontrolled systemic infection requiring hospitalization.
* Immunocompromised participants with increased risk of opportunistic infections, including known human immunodeficiency virus (HIV)-positive participants with cluster of differentiation 4 (CD4) counts ≤350 cells/millimeters (mm^3) or history of opportunistic infection in the last 12 months.
* Participants with a known active or chronic hepatitis B or active hepatitis C virus (HCV) infection. Participants with a history of HCV infection who have completed curative therapy for HCV at least 12 weeks before the Screening Visit and have a documented undetectable viral load at the Screening Visit are eligible for enrollment.
* Participants who have not adequately recovered from a major surgery within 4 weeks of starting study drug administration.
* Participants who received any other investigational agents within 4 weeks of the Screening Visit or <5 half-lives since completion of previous investigational therapy have elapsed, whichever is shorter.
* Participants who have a hypersensitivity to arsenic.
* Participants who have experienced the following Grade ≥3 non-hematologic toxicities associated with ATO administration: QT prolongation, hepatotoxicity, neurotoxicity, cardiac function abnormalities. Participants who experienced other severe and life-threatening clinically-significant ATO-related AEs that are considered, in the judgement of the investigator, to increase participant risk with continued ATO treatment are also excluded.

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Single-Dose Module: Maximum Observed Plasma Concentration (Cmax) of SY-2101 | Predose and up to 168 hours postdose
Single-Dose Module: Area Under the Curve (AUC) of SY-2101 | Predose and up to 168 hours postdose
Multiple-Dose Module: Cmax of SY-2101 | Predose and up to 6 hours postdose on Day 5 and up to 4 hours postdose on Day 26
Multiple-Dose Module: AUC of SY-2101 | Predose and up to 6 hours postdose on Day 5 and up to 4 hours postdose on Day 26

SECONDARY OUTCOMES:
Single-Dose Module: Cmax of ATO | Predose and up to 168 hours postdose
Single-Dose Module: AUC of ATO | Predose and up to 168 hours postdose
Multiple-Dose Module: Cmax of ATO | Predose and up to 6 hours postdose on Day 5 and up to 4 hours postdose on Day 26
Multiple-Dose Module: AUC of ATO | Predose and up to 6 hours postdose on Day 5 and up to 4 hours postdose on Day 26
Number of Participants With Adverse Events | up to Day 23 for single-dose module and up to Day 56 for multiple-dose module

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Syros Pharmaceuticals Inc.
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern Memorial Hospital, Chicago, Illinois
  - John Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Weill Cornell Medical College, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ravandi F, Rangaraju S, Kantarjian H, Garcia-Manero G, Yilmaz M, Baker K, Hall T, Grabenstein J, Roy P, Zamboni BA, Zamboni WC, Warlick E, Kelly M, Roth DA, Ghiaur G. A pharmacokinetic and safety study of oral arsenic trioxide in patients with acute promyelocytic leukemia. Blood Adv. 2025 May 13;9(9):2136-2143. doi: 10.1182/bloodadvances.2024015453. PMID 40020161